CLINICAL TRIAL: NCT02299934
Title: 3T MR Angiography of the Hepatic Vasculature: A Pilot Comparison Study of New Noncontrast Techniques to Post-contrast Technique and CT Angiography in Liver Donors.
Brief Title: 3T MR Angiography of the Hepatic Vasculature
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of support
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-1213
Record Dates: First submitted 2014-11-14; First posted 2014-11-24 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Liver Blood Supply
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects who fulfill the criteria for living liver donation (Other): Subjects who fulfill the criteria for living liver donation and are evaluated for the procedure with Computerized Tomography (CT) and Magnetic Resonance Imaging (MRI).
  Interventions: Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: Compurtized Tomgraphy (CT)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — MRI sequences for visualisation of the blood supply of liver without contrast agent.
Diagnostic Test: Compurtized Tomgraphy (CT) — CT including CT Angiography (CTA) for the evaluation of hepatic vasculature.

SUMMARY:
This study plans to learn more about the two Magnetic Resonance Angiography (MRA) techniques.

DETAILED DESCRIPTION:
This study will use two Magnetic Resonance Angiography (MRA) techniques that will look at participants liver veins and arteries without giving a coloring matter (contrast) before taking the images. Investigators propose to evaluate the usefulness of these two new techniques, which do not involve exposing participants to radiation or contrast.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that fulfill the criteria for living liver donation and are evaluated for the procedure with CT and MR.

Exclusion Criteria:

* Unable to give informed consent
* Unable to comply with breathing or other imaging related instructions resulting in inability to obtain diagnostic quality MRI studies
* Not suitable to undergo MRI with a gadolinium-based contrast agent because of:

  * Claustrophobia, unless patient agrees to sedation measures per institutional standard practice during MR imaging
  * Presence of metallic objects or implanted medical devices in body per institutional safety standards
  * Weight greater than that allowable by the MR table
  * Renal failure, as determined by estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 by the Modification of Diet in Renal Disease (MDRD) model based on a serum creatinine level obtained within 28 days prior to enrollment
  * Known allergy-like reaction to contrast media (gadolinium) or moderate or severe allergic reactions to one or more allergens as defined by the American College of Radiology (ACR), and unwillingness to undergo pre-treatment as defined by the institution's policy and/or ACR guidance
  * Pregnancy (if a female is of childbearing potential --defined as a premenopausal female capable of becoming pregnant --a pregnancy test should be done)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-07; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Chang, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No
Participant data will only be shared to research personnel.

REFERENCES:
- [Background] Puippe GD, Alkadhi H, Hunziker R, Nanz D, Pfammatter T, Baumueller S. Performance of unenhanced respiratory-gated 3D SSFP MRA to depict hepatic and visceral artery anatomy and variants. Eur J Radiol. 2012 Aug;81(8):e823-9. doi: 10.1016/j.ejrad.2012.02.016. Epub 2012 May 10. PMID 22578837

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects Who Fulfill the Criteria for Living Liver Donation
Started | 13
Completed | 0
Not Completed | 13
Not completed — Termination of study | 13

BASELINE CHARACTERISTICS:
Population: 13 patients were consented and began the preliminary examination. 11 completed the preliminary examination after consenting.
Arm/Group | Subjects Who Fulfill the Criteria for Living Liver Donation
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Liver Blood Supply Diameters
Time Frame: Day 1
Population: Study was terminated prior to collecting any outcome measure data.
Arm/Group | Subjects Who Fulfill the Criteria for Living Liver Donation
Number analyzed (Participants) | 0

2. Primary Outcome: The Visibility of the Variations of the Liver Blood Supply
Time Frame: Day 1
Population: Study was terminated prior to collecting any outcome measure data.
Arm/Group | Subjects Who Fulfill the Criteria for Living Liver Donation
Number analyzed (Participants) | 0

3. Primary Outcome: Detection Rates of the Variations of the Liver Blood Supply
Time Frame: Day 1
Population: Study was terminated prior to collecting any outcome measure data.
Arm/Group | Subjects Who Fulfill the Criteria for Living Liver Donation
Number analyzed (Participants) | 0

4. Primary Outcome: The Percentage of Examinations With the Presence of Significant Artifacts Interfering Interpretation.
Time Frame: Day 1
Population: Study was terminated prior to collecting any outcome measure data.
Arm/Group | Subjects Who Fulfill the Criteria for Living Liver Donation
Number analyzed (Participants) | 0

5. Primary Outcome: How Badly the Artifacts Prevented Evaluation by the Reader.
Time Frame: Day 1
Population: Study was terminated prior to collecting any outcome measure data.
Arm/Group | Subjects Who Fulfill the Criteria for Living Liver Donation
Number analyzed (Participants) | 0

6. Primary Outcome: The Relative Signal Intensity of the Liver Blood Supply
Time Frame: Day 1
Population: Study was terminated prior to collecting any outcome measure data.
Arm/Group | Subjects Who Fulfill the Criteria for Living Liver Donation
Number analyzed (Participants) | 0

7. Primary Outcome: Documentation of Acquisition Time
Time Frame: Day 1
Population: Study was terminated prior to collecting any outcome measure data.
Arm/Group | Subjects Who Fulfill the Criteria for Living Liver Donation
Number analyzed (Participants) | 0

8. Secondary Outcome: The Percentage of Examinations That Caused Adverse Events
Time Frame: Day 1
Population: Study was terminated prior to collecting any outcome measure data.
Arm/Group | Subjects Who Fulfill the Criteria for Living Liver Donation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Duration of study activity (approximately 2 years)
Description: This study was terminated early due to lack of enrollment. No adverse events data was reported prior to early termination
Arm/Group | Subjects Who Fulfill the Criteria for Living Liver Donation
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

LIMITATIONS AND CAVEATS:
Study was terminated prior to collecting any outcome measure data or performing any image analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT02299934/Prot_SAP_000.pdf